CLINICAL TRIAL: NCT07086170
Title: The Effect of Psychological First Aid Training on Disaster Response Self-Efficacy: A Randomized Controlled Study
Brief Title: Psychological First Aid Training for Nursing Students
Acronym: PFA-EDU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nurhayat Kiliç Bayageldi (Other)
Responsible Party: Sponsor-Investigator, Nurhayat Kiliç Bayageldi, Assistant Professor, Artvin Coruh University
Organization: Artvin Coruh University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: E-18457941-050.99-50732
Record Dates: First submitted 2025-07-18; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Emergency Preparedness; Nursing Students; Crisis Intervention; Self-Efficacy
Keywords: Disaster; psychological first aid; nursing students; randomized controlled trial

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial was conducted according to the CONSORT guideline.
Masking Description: Open-label design; no blinding was used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): This group received online psychological first aid (PFA) training. Students were randomly divided into four subgroups. Each group received six 60-minute sessions over three weeks. Sessions included slides, videos, Q&A, role-plays, and case-based discussions. Group members shared thoughts, asked questions, and practiced PFA scenarios. A 17-minute PFA video was also shown. The training was delivered by the researcher and emphasized core PFA principles such as safety, calmness, and self-efficacy.
  Interventions: Other: Psychological First Aid Training
- Control Group (No Intervention): Participants in this group did not receive any training during the study period. They continued with their standard nursing curriculum without any additional intervention.

INTERVENTIONS:
Other: Psychological First Aid Training — Structured training based on psychological first aid principles. Delivered in six 60-minute sessions over three weeks. Includes theoretical content, interactive methods, and case-based exercises to build disaster response competencies.
  Other Names: PFA Training
  Arms: Intervention Group

SUMMARY:
This randomized controlled trial aimed to evaluate the effect of psychological first aid (PFA) training on disaster response and psychological first aid application self-efficacy among nursing students. The study included 132 participants, with 72 in the intervention group and 60 in the control group. The intervention group received six 60-minute online PFA training sessions over three weeks. Data were collected using the Personal Information Form, Disaster Response Self-Efficacy Scale (DRSES), and the Psychological First Aid Application Self-Efficacy Scale. After the training and follow-up, the intervention group showed significantly higher self-efficacy scores across all DRSES sub-dimensions and in applying PFA, compared to the control group. Findings suggest that integrating PFA training into nursing education can enhance students' readiness and competence in disaster response.

DETAILED DESCRIPTION:
Disasters pose significant challenges to healthcare systems and frontline professionals, particularly nurses. Psychological first aid (PFA) is a fundamental psychosocial support approach that aims to reduce stress, promote adaptive functioning, and improve psychological well-being in individuals affected by disasters. However, nursing students often lack formal training in disaster preparedness and psychosocial interventions.

This randomized controlled trial was conducted to evaluate the effect of psychological first aid training on disaster response self-efficacy and psychological first aid application self-efficacy among senior nursing students. The study was designed according to the CONSORT guidelines and included a total of 132 participants, with 72 students in the intervention group and 60 in the control group. Students in the intervention group received a total of six 60-minute online PFA training sessions delivered twice a week for three weeks. The training content was based on internationally recognized PFA principles.

Data collection tools included the Personal Information Form, the Disaster Response Self-Efficacy Scale (DRSES), and the Psychological First Aid Application Self-Efficacy Scale. Measurements were taken before the training, immediately after the training, and at 3 months follow-up. Results showed significant improvements in the intervention group's scores across all sub-dimensions of disaster response self-efficacy (on-site rescue competency, disaster psychological nursing competency, quality of role undertaken, and adaptation competency) and in their perceived self-efficacy to apply PFA, compared to the control group.

These findings emphasize the importance of integrating structured PFA training into nursing education to enhance disaster preparedness and psychosocial intervention competencies among future healthcare professionals.

ELIGIBILITY:
Inclusion Criteria:Volunteered to participate after being informed about the study

Were fourth-year nursing students at the participating universities

Had not previously participated in similar training that could bias results

Had not received any prior psychological first aid (PFA) training or services

Had no internet access problems during the intervention period -

Exclusion Criteria:Individuals who did not complete the post-training or follow-up assessments

Students who withdrew from the study voluntarily during the intervention process

Participants who experienced technical issues that prevented their attendance in most training sessions

Individuals with prior experience in psychological first aid or formal training in disaster response

-

Ages: 21 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2023-04-02 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Disaster Response Self-Efficacy Scale | aseline, post-intervention (Week 3), and follow-up (Month 3)
  Developed by Hong-Yan Li et al. (2017), this scale assesses individuals' perceived self-efficacy in effectively responding to disasters. The Turkish adaptation, including validity and reliability studies, was conducted by Koca et al. (2018). The scale consists of 19 items across three sub-dimensions, rated on a five-point Likert scale ranging from 1 (No self-confidence) to 5 (Full self-confidence). Higher total scores reflect greater self-efficacy in disaster response. The original study reported excellent internal consistency, with a Cronbach's alpha of 0.96 for the overall scale, and 0.93 for each sub-dimension: On-site Rescue Competence, Psychological Nursing Competence in Disaster, and Quality of Role Undertaken in Disaster and Adaptation Competence.21 In the present study, Cronbach's alpha values ranged from 0.87 to 0.93 across groups and time points, confirming the scale's reliability in this sample
Psychological First Aid Application Self-Efficacy Scale | aseline, post-intervention (Week 3), and follow-up (Month 3)
  Developed by Kılıç Bayageldi and Şimşek (2022), this scale assesses self-efficacy in applying Psychological First Aid (PFA). It consists of 35 items within a single sub-dimension, rated on a five-point Likert scale from 1 (Not at all appropriate) to 5 (Completely appropriate). Total scores range from 35 to 175, with no reverse-scored items. Higher scores indicate greater self-efficacy in PFA application. The scale demonstrated excellent reliability, with a Cronbach's alpha of 0.95 and a test-retest correlation coefficient of 0.93.22 In this study, internal consistency remained high across all measurements, with Cronbach's alpha values between 0.89 and 0.96.

CONTACTS AND LOCATIONS:
Overall Officials: Nurhayat KILIÇ BAYAGELDİ, PhD, Principal Investigator — Artvin Coruh University
Locations (1):
- Artvin Coruh University, Artvin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No